CLINICAL TRIAL: NCT02083224
Title: Familial Cancer Registry and DNA Bank
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Lee Soo Chin, National University Hospital, Singapore
Other Study IDs: 2000/00511
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood for DNA banking and future genotyping Questionnaires regarding family history of cancer and personal medical history will be taken.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cancer patients

SUMMARY:
Clinical cancer genetics is an emerging new field in medical oncology, and has been incorporated into routine oncology practice in many leading medical institutions in North America and Europe. Cancer genetics is the study of genetic factors contributing to carcinogenesis. In the last 5-10 years, genes responsible for various well-defined hereditary cancer syndromes have been cloned. These include the BRCAJ/2 genes in hereditary breast and ovarian cancer syndrome, the A4PC gene in Familial Adenomatous Polyposis, and the mismatch repair genes (hMLH1, hMSH2, hPMS1, hPMS2, hMSH6) in hereditary non-polyposis colorectal cancer (HNPCC). One of the goals of a clinical cancer genetics service is to identify families at risk for hereditary cancer syndromes, provide genetic counseling, and offer genetic testing when appropriate. The identification of causative genes in hereditary cancer syndromes together with the advent of genetic testing is starting to have an impact on clinical management. The ability to identify a gene mutation in a cancer family allows predictive testing, stratifying at-risk family members into carriers who will benefit from aggressive surveillance and/or preventive options, and non-carriers who may be spared unnecessary surveillance. Appropriate use of genetic testing will ultimately result in medical cost reduction.

The investigators hypothesize that the clinical characteristics and genetic factors contributing to hereditary cancer in the Singaporean Asian population are distinct from those described for Western patients.

ELIGIBILITY:
Inclusion Criteria:

* Any individual with very early onset cancer (eg diagnosed before age 40).
* Any family with three or more first- or second-degree relatives with the same cancer
* Any individual with two or more different primary cancers
* Any family that fulfils diagnostic criteria for known hereditary cancer syndromes

Exclusion Criteria:

Nil

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are recruited from the National University Hospital. All cancer patients seen in the Cancer Centre, NUH, are screened using a basic family history form.The family history is reviewed by the Principal Investigator with the cancer genetics counselor. Eligible patients who fulfil the eligibility criteria as described below are invited to participate. Written informed consent is obtained. Demographic characteristics and cancer history of the study subject is prospectively recorded. Participants are invited to fill out a family history questionnaire providing cancer history information on their first- and second-degree relatives. Participants are also invited to donate 10ml blood for DNA banking and future genotyping. Permission will be obtained from participants to contact family members who may be eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2000-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in genetics testing method | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Petersen GM, Brensinger JD, Johnson KA, Giardiello FM. Genetic testing and counseling for hereditary forms of colorectal cancer. Cancer. 1999 Dec 1;86(11 Suppl):2540-50. doi: 10.1002/(sici)1097-0142(19991201)86:11+3.0.co;2-8. PMID 10630180
- [Background] Giardiello FM, Brensinger JD, Petersen GM, Luce MC, Hylind LM, Bacon JA, Booker SV, Parker RD, Hamilton SR. The use and interpretation of commercial APC gene testing for familial adenomatous polyposis. N Engl J Med. 1997 Mar 20;336(12):823-7. doi: 10.1056/NEJM199703203361202. PMID 9062090